CLINICAL TRIAL: NCT02696122
Title: Quality of Recovery After Local Infiltration Under General Anesthesia Via Laryngeal Mask or Spinal Anesthesia for Inguinal Hernia Repair.
Brief Title: Quality of Recovery After General or Spinal Anesthesia for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUCSP 1.316.318
Record Dates: First submitted 2016-02-23; First posted 2016-03-02 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Quality of Life; Pain, Postoperative; Personal Satisfaction; Postoperative Complication
Keywords: Pain, postoperative; Hernia, abdominal; Anesthesia, spinal; Anesthesia, local; Anesthesia, general; Quality of life; Anesthesia recovery period; Personal satisfaction; Postoperative complications; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction; Postoperative Complications; Hernia, Abdominal | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Group (Experimental): Local infiltration under general anesthesia via laryngeal mask
  Interventions: Procedure: Local Group
- Spinal Group (Experimental): Spinal anesthesia with 15 mg of 0.5% hyperbaric bupivacaine
  Interventions: Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: Local Group — General anesthesia willl be induced with propofol 2 mg mg. kg-1 and alfentanyl 30 mcg.kg-1. Once an appropriate depth of anesthesia had been obtained, a laryngeal mask airway (LMA) will be positioned. The anesthesia will be maintained by propofol 4 to 5 mg. kg-1.h-1. Ventilation will controlled by adjusting the flow volume and respiratory rate to keep the end-tidal CO2 level (PETCO2) between 30 and 40 mmHg. For local anesthesia, approximately 50 ml of 0.5% ropivacaive will infiltrated along the line of incision in the subcutaneous plane, followed by peripheral nerve block technique (e.g., ilioinguinal-hypogastric nerve block) and local wound infiltration at the fascial level.
  Other Names: Local anesthesia under general anesthesia via laryngeal mask
  Arms: Local Group
Procedure: Spinal anesthesia — Spinal puncture will be performed with the patient in the sitting position, using 27G disposable Quincke needles (B. Braun, Meisungen, AG). After obtaining CSF, 15 mg of 0.5% hyperbaric bupivacaine will be injected.
  Arms: Spinal Group

SUMMARY:
Different anesthetic techniques have been proposed for carrying out Inguinal hernia repair, including local anesthesia, regional and general. There are no recent data on the application of a validated questionnaire to assess which anesthetic technique, local infiltration under general anesthesia or spinal anesthesia, would provide better quality of recovery in the opinion of the patients undergoing inguinal hernia repair. The aim of the study is to perform a randomized clinical trial comparing the quality of recovery (QoR-40) after local infiltration under general anesthesia via laryngeal mask (LMA) or spinal anesthesia for unilateral inguinal hernia repair. METHODS - Seventy patients aged 18 to 65 years old, who were scheduled to undergo unilateral inguinal hernia repair at Santa Lucinda Hospital will be enrolled in the study. The anesthesia will be performed according to the following sequence: L Group - intravenous (I.V.) propofol and alfentanyl, followed by LMA positioning. The anesthesia will be maintained by propofol. For local anesthesia, approximately 50 ml of 0.5% ropivacaine will be infiltrated along the line of incision in the subcutaneous plane, followed by peripheral nerve block technique (e.g., ilioinguinal-hypogastric nerve block) and local wound infiltration at the fascial level. S Group - spinal puncture followed by intrathecal 15 mg of 0.5% hyperbaric bupivacaine injection and sedation with propofol by continuous infusion. Pain will be assessed every 15 minutes at Post-anesthesia Care Unit (PACU) using a 0-10 numeric pain rating scale and I.V. morphine will be administered to maintain the pain score below 4. The QoR-40 will be administered by a blind investigator 24 hours after surgery.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most commonly performed operations worldwide. The recommended treatment is surgery, which has undergone important advances in the last two decades. Different anesthetic techniques have been proposed for carrying out such procedures, including local anesthesia, regional and general. Even though local anesthesia (so called monitored anesthesia care) is a more cost effective anesthetic technique for inguinal hernia repair, general and spinal anesthesia remain the most popular anesthetic techniques at university based teaching programs. It has been suggested that the use of local anesthetic techniques requires greater surgical skill in the handling of tissues and that, therefore, less skilled surgeons find it more convenient to operate under general or spinal anesthesia. The choice of anesthesia is influenced by several factors, including surgeon or anesthesiologist preferences, patient characteristics, cost or length of hospital stay. Despite its popularity, spinal anesthesia can lead to side effects as urinary retention, hypotension, motor block of lower extremities and headache. A recent systematic review evaluated studies on the influence of anesthetic technique in controlling the occurrence of postoperative pain in patients undergoing inguinal hernia repair. According to the authors, local anesthesia, with or without general anesthesia is more effective considering the avoidance of adverse events compared to spinal anesthesia. Traditionally, anesthesia and surgery studies have assessed outcomes such as time to wake or hospital stay and the incidence of nausea, vomiting, pain or other adverse events. Recently, a measurement that probes quality of life from the perspective of the patient has been considered as a more important factor in clinical studies that wish to investigate the effect of anesthesia and surgery on patient recovery and satisfaction. The Quality of Recovery-40 questionnaire (QoR-40), a validated instrument for this purpose, allows an objective evaluation of the factors that can influence the perception of the patient, and has been used successfully to assess the degree of recovery after several different surgical and anesthetic techniques. There are no recent data on the application of this instrument to assess which anesthetic technique, local infiltration under general anesthesia via laryngeal mask or spinal anesthesia, would provide better quality of recovery in the opinion of the patients undergoing inguinal hernia repair. The aim of the study is to perform a randomized clinical trial comparing the quality of recovery after local infiltration under general anesthesia via laryngeal mask or spinal anesthesia for unilateral inguinal hernia repair.

METHODS This randomized trial was approved by the Research Ethics Committee of the School of Medical and Health Sciences, Pontifical Catholica University of São Paulo, approval number 45087615.0.0000.5373. Written consent form will be obtained from all participants. Seventy patients aged 18 to 65 years old, with an American Society of Anesthesiologists (ASA) physical status I or II, who will bee scheduled to undergo local infiltration under general anesthesia via laryngeal mask or spinal anesthesia for unilateral inguinal hernia repair at Santa Lucinda Hospital will be enrolled in the study. Patients who (i) refuse to participate in the study; (ii) are not able to communicate due to alterations in the level of consciousness, or neurologic, or psychiatric disease; (iii) present with contraindication to any of the drugs used in the present study; (iv) have history of alcohol or drug dependence; (v) are super obese as defined by a body mass index (BMI) ≥ 40; and (vi) undergo operation for recurrent, strangulated, incarcerated or bilateral hernia will excluded from the study.

Study Sequence No premedication will be applied to the patients. Patients´ preoperative data including age, gender, physical status, BMI and hernia type according to Nyhus classification will be collected

Randomization The sample size for the following step was calculated considering 90% power to detect a 10-point difference in QoR-40, which indicated the need to include 31 participants in each group. Taking possible losses into consideration, the final sample will include 70 participants, which will be allocated to two groups according to a random number sequence from a web-based random-number generator (available at www.random.com). Because of significant difference between the anesthetic techniques, the patient and the investigators will be blinded to group allocation, but not the anesthesia. The anesthetic technique to be used for each individual participant will be kept in an opaque and sealed envelope, which will be opened at the time of surgery.

Anesthesia

On arrival at the operating room, standard ASA monitors will be applied. Intravenous midazolam (0.06 to 0.08 mg.kg-1) and 1% lidocaine (30 mg) will be administered immediately after venoclysis. The anesthesia will be performed according to the following sequence:

L Group - General anesthesia willl be induced with propofol 2 mg mg. kg-1 and alfentanyl 30 mcg.kg-1. Once an appropriate depth of anesthesia had been obtained, a laryngeal mask airway (LMA) will be positioned. The anesthesia will be maintained by propofol 4 to 5 mg. kg-1.h-1. Ventilation will be controlled by adjusting the flow volume and respiratory rate to keep the end-tidal CO2 level (PETCO2) between 30 and 40 mmHg. For local anesthesia, approximately 50 ml of 0.5% ropivacaine will be infiltrated along the line of incision in the subcutaneous plane, followed by peripheral nerve block technique (e.g., ilioinguinal-hypogastric nerve block) and local wound infiltration at the fascial level. Failure of local anesthesia will be defined as the presence of movements, sweating, tachycardia or blood pressure increase >10% of the pre-induction value with the beginning of the surgery. In these cases further infiltration of additional 10 mL of 0.5% ropivacaine will be allowed. At the end of the surgery, propofol will be discontinued and the LMA removed whenever the patients resume adequate spontaneous breathing.

S Group - In the S group, spinal puncture will be performed with the patient in the sitting position, using 27 Gauge (27G) disposable Quincke needles (B. Braun, Meisungen, AG). After obtaining cerebral spinal fluid (CSF), 15 mg of 0.5% hyperbaric bupivacaine will be injected. In case of complete failure, a new puncture will be performed and the same dose of anesthetic drug injected. In cases of partial failure, the anesthesia will be converted to general anesthesia and the patient excluded from the study. All the patients will be sedated with propofol by continuous infusion at an initial dose of 0.5 mg.kg-1 followed by 2 to 5 mg. kg-1.h-1 as necessary to reach level 5 on Ramsay Sedation Scale. The Lichtenstein tension-free method of inguinal hernia repair will be used in both groups and all procedures will be performed by the same surgical team. Patients who exhibit reductions in systolic arterial pressure (SAP) greater than 30% will be given ephedrine (10 mg). Lactated Ringer's solution will be used for fluid replacement therapy at a rate of approximately 500 ml throughout the first 30 minutes, and, then, 2 ml.kg-1.h-1. All of the participants will be given i.v. ketoprofen (100 mg) before the end of the surgery. The time to operating room discharge will be registered.

Postoperative When stable vital signs and respiration was confirmed, all patients will be transferred to the post-anesthesia care unit (PACU). Data related to the occurrence of pain, nausea, vomiting, shivering, urinary retention and the length of stay at the PACU will be recorded. Pain will be assessed every 15 minutes using a 0-10 numeric pain rating scale, where zero meant no pain and 10 the worst imaginable pain. Intravenous morphine (1 to 2 mg) will be administered every 15 minutes to maintain the pain score below 4 (1 mg when the pain score was <7 and 2 mg when it was ≥7). Postoperative pain relief in the ward was accomplished by i.v. ketoprofen (100 mg) every 12 hours, dipyrone (30 mg.kg-1, maximum 1 g) every six hours and tramadol (100 mg) at eight-hour minimum intervals as needed whenever patients judge that their analgesia is insufficient. Postoperative nausea and vomiting (PONV) will be treated with i.v. dimenhydrinate (30 mg). Pain score, use of analgesics, and the occurrence of nausea, vomiting, and other complications during the hospital ward stay will be recorded.

QoR-40 Questionnaire The quality of postoperative functional recovery will be assessed by the QoR-40 questionnaire, which assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item was rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II , who will be scheduled to undergo unilateral inguinal hernia repair

Exclusion Criteria:

* Patients who (i) refuse to participate in the study; (ii) are not able to communicate due to alterations in the level of consciousness, or neurologic, or psychiatric disease; (iii) present with contraindication to any of the drugs used in the present study; (iv) have history of alcohol or drug dependence; (v) are super obese as defined by a body mass index (BMI) ≥ 40; and (vi) undergo operation for recurrent, strangulated, incarcerated or bilateral hernia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Quality of recovery from anesthesia | 24 hours
  The quality of postoperative functional recovery will be assessed by the QoR-40 questionnaire, which assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item was rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  Pain will be assessed every 15 minutes using a 0-10 numeric pain rating scale, where zero meant no pain and 10 the worst imaginable pain. Intravenous morphine (1 to 2 mg) will be administered every 15 minutes to maintain the pain score below 4 (1 mg when the pain score was <7 and 2 mg when it was ≥7). Postoperative pain relief in the ward was accomplished by i.v. ketoprofen (100 mg) every 12 hours, dipyrone (30 mg.kg-1, maximum 1 g) every six hours and tramadol (100 mg) at eight-hour minimum intervals as needed whenever patients judge that their analgesia is insufficient.
Adverse events | 24 hours
  Occurrence of nausea, vomiting, shivering, urinary retention

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, PhD, Principal Investigator — School of Medical and Health Sciences, Pontificial Catholic University of São Paulo
Locations (1):
- Santa Lucinda Hospital, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kehlet H, White PF. Optimizing anesthesia for inguinal herniorrhaphy: general, regional, or local anesthesia? Anesth Analg. 2001 Dec;93(6):1367-9. doi: 10.1097/00000539-200112000-00001. No abstract available. PMID 11726407
- [Background] Nordin P, Zetterstrom H, Gunnarsson U, Nilsson E. Local, regional, or general anaesthesia in groin hernia repair: multicentre randomised trial. Lancet. 2003 Sep 13;362(9387):853-8. doi: 10.1016/S0140-6736(03)14339-5. PMID 13678971
- [Background] O'Dwyer PJ, Serpell MG, Millar K, Paterson C, Young D, Hair A, Courtney CA, Horgan P, Kumar S, Walker A, Ford I. Local or general anesthesia for open hernia repair: a randomized trial. Ann Surg. 2003 Apr;237(4):574-9. doi: 10.1097/01.SLA.0000059992.76731.64. PMID 12677155
- [Background] Bakota B, Kopljar M, Baranovic S, Miletic M, Marinovic M, Vidovic D. Should we abandon regional anesthesia in open inguinal hernia repair in adults? Eur J Med Res. 2015 Sep 17;20(1):76. doi: 10.1186/s40001-015-0170-0. PMID 26381501
- [Background] Joshi GP, Rawal N, Kehlet H; PROSPECT collaboration; Bonnet F, Camu F, Fischer HB, Neugebauer EA, Schug SA, Simanski CJ. Evidence-based management of postoperative pain in adults undergoing open inguinal hernia surgery. Br J Surg. 2012 Feb;99(2):168-85. doi: 10.1002/bjs.7660. Epub 2011 Sep 16. PMID 21928388
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540

DOCUMENTS (2):
  • Study Protocol (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT02696122/Prot_000.pdf
  • Informed Consent Form (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT02696122/ICF_001.pdf